CLINICAL TRIAL: NCT04975542
Title: Efficacy of Osteopathic Manipulation on Breathing Mechanics in a Healthy Population: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jayla Bostic (Other)
Responsible Party: Sponsor-Investigator, Jayla Bostic, Medical Student, The Touro College and University System
Organization: The Touro College and University System (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T2022
Record Dates: First submitted 2021-05-19; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Respiratory Function Impaired
Keywords: Breathing Mechanics; Osteopathic Manipulative Treatment; Chest Wall Excursion; Pulmonary Function Tests
MeSH Terms: conditions — Respiratory Insufficiency | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Other: Osteopathic Manipulative Medicine
- Sham Group (Sham Comparator)
  Interventions: Other: Sham

INTERVENTIONS:
Other: Osteopathic Manipulative Medicine — Manipulative therapies based on Osteopathic principles.
  Arms: Treatment Group
Other: Sham — Light touch techniques to mimic to osteopathic treatment.
  Arms: Sham Group

SUMMARY:
This study focused on improving breathing mechanics by using various osteopathic manipulative therapy (OMT) techniques. The investigators randomly assigned participants to a control group who received sham treatment and a treatment group who received OMT. The investigators measured variable pre- and post- treatment on both groups. The investigators observed an improvement in breathing mechanics in the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers from Touro College of Osteopathic Medicine (TouroCOM), including students and staff, were recruited as subjects of this study. Any participant with recent or past medical history of obstructive or restrictive lung disorders, recent trauma, or illnesses, and/or chest abnormalities were excluded from the study.

Exclusion Criteria:

* Certain study results were excluded on the basis of abnormal baseline measurements, including but not limited to, heart rate, oxygen saturation, respiratory rate, improper spirometer use, technique and/or high variance among the repeated measurements obtained for each participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Change in chest wall excursion | Measure assessing a change from baseline chest wall excursion within 5 minutes of treatment completion.
  M1 and M2 measurements with a soft tape measure. M1: Level of sternal notch (in centimeters), M2: Level of xiphoid process (in centimeters).
Change in forced vital capacity (FVC) | Measure assessing a change from baseline FVC value via pulmonary function testing within 5 minutes of treatment completion.
  Measurement of Forced Vital Capacity (FVC) as measured via pulmonary function testing.
Change in forced expiratory volume at 1 second (FEV1) | Measure assessing a change from baseline in forced expiratory volume at 1 second via pulmonary function testing within 5 minutes of treatment completion.
  Measurement of Forced Expiratory Volume at 1 second (FEV1) as measured via pulmonary function testing.
Change in FEV1/FVC ratio | Measure assessing a change from baseline FEV1/FVC ratio value via pulmonary function testing within 5 minutes of treatment completion.
  Measurement of a ratio between FEV1 and FVC values that are obtained through pulmonary function testing.

SECONDARY OUTCOMES:
Change in respiratory rate | Measure assessing a change from baseline respiratory rate within 5 minutes of treatment completion.
  Measurement with a timer-based breath count with the units of breaths per minute.
Change in heart rate | Measure assessing a change from baseline heart rate within 5 minutes of treatment completion.
  Measurement with a noninvasive finger pulse-oximeter device with the units of beats per minute (bpm).
Oxygen Saturation (spO2) | Measure assessing a change from baseline oxygen saturation within 5 minutes of treatment completion.
  Measurement with a noninvasive finger pulse-oximeter with the unit of spO2.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Volokitin, MD, DO, Study Director — Touro College of Osteopathic Medicine
Locations (1):
- Touro College of Osteopathic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noll DR, Degenhardt BF, Stuart M, McGovern R, Matteson M. Effectiveness of a sham protocol and adverse effects in a clinical trial of osteopathic manipulative treatment in nursing home patients. J Am Osteopath Assoc. 2004 Mar;104(3):107-13. No abstract available. PMID 15083985
- [Background] Zanotti E, Berardinelli P, Bizzarri C, Civardi A, Manstretta A, Rossetti S, Fracchia C. Osteopathic manipulative treatment effectiveness in severe chronic obstructive pulmonary disease: a pilot study. Complement Ther Med. 2012 Feb-Apr;20(1-2):16-22. doi: 10.1016/j.ctim.2011.10.008. Epub 2011 Nov 27. PMID 22305244
- [Background] Guiney PA, Chou R, Vianna A, Lovenheim J. Effects of osteopathic manipulative treatment on pediatric patients with asthma: a randomized controlled trial. J Am Osteopath Assoc. 2005 Jan;105(1):7-12. PMID 15710659
- [Background] Kaneko H, Shiranita S, Horie J, Hayashi S. Reduced Chest and Abdominal Wall Mobility and Their Relationship to Lung Function, Respiratory Muscle Strength, and Exercise Tolerance in Subjects With COPD. Respir Care. 2016 Nov;61(11):1472-1480. doi: 10.4187/respcare.04742. Epub 2016 Oct 18. PMID 27794081
- [Background] Lorenzo S, Nicotra CM, Mentreddy AR, Padia HJ, Stewart DO, Hussein MO, Quinn TA. Assessment of Pulmonary Function After Osteopathic Manipulative Treatment vs Standard Pulmonary Rehabilitation in a Healthy Population. J Am Osteopath Assoc. 2019 Feb 11. doi: 10.7556/jaoa.2019.026. Online ahead of print. PMID 30741314